CLINICAL TRIAL: NCT05519137
Title: Using a Wireless Controller to Deliver a Lighting Intervention to Persons With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Mariana Figueiro, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY-20-01772
Record Dates: First submitted 2022-08-25; First posted 2022-08-29 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Participants will randomly be assigned to initially receive the active or control lighting intervention
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active lighting intervention then Control lighting condition (Active Comparator): Each lighting condition will be 8 weeks in length. After a 4 week washout, each participant will crossover to the opposite condition.
  Interventions: Device: Active lighting intervention; Device: Control lighting intervention
- Control lighting condition then Active light intervention (Active Comparator): Each lighting condition will be 8 weeks in length. After a 4 week washout, each participant will crossover to the opposite condition.
  Interventions: Device: Active lighting intervention; Device: Control lighting intervention

INTERVENTIONS:
Device: Active lighting intervention — Lighting intervention designed to impact the circadian system
Device: Control lighting intervention — Lighting intervention designed to have no impact on the circadian system

SUMMARY:
To test the effect of a tailored lighting intervention controlled by the Readings At Desk (RAD) controller on sleep and mood in Alzheimer's disease participants.

DETAILED DESCRIPTION:
Each participant will be enrolled for 22 weeks. Participants will be randomly assigned to receive either the active or control lighting condition. Each lighting condition will be 8 weeks in length. After a 4 week washout, each participant will crossover to the opposite condition. Assessments will be performed before and at the end of each lighting intervention.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of Alzheimer's disease with a Mini Mental Score Examination (MMSE) between 0 and 19
* a score >5 on the PSQI.

Exclusion criteria:

- use of sleep medication

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Sleep disturbance using the Pittsburgh Sleep Quality Index | up to 22 weeks
  The Pittsburgh Sleep Quality Index (PSQI) is composed of 19 items that generate 7 component scores. The sum of the 7 component scores yields a single global score with a range of 0 to 21. A global score >5 is considered to indicate sleep disturbances. A lower global score indicates improvement in sleep disturbance.

SECONDARY OUTCOMES:
Depression screening utilizing the Cornell Scale for Depression in Dementia (CSDD) | up to 22 weeks
  The CSDD is a a 19-item tool designed to rate symptoms of depression in patients with dementia. This tool evaluates the presence and extent of mood-related signs. Scores range from 0 to 38 with a higher score indicating higher depressive symptoms.
Sleep efficiency measured by actigraphy | up to 22 weeks
  Sleep efficiency is calculated from the wrist worn actigraph by the software program as the percentage of the time in bed spent sleeping. The ratio of total sleep time (TST) to total time in bed (TIB) multiplied by 100 to yield a percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Mariana Figueiro, PhD, Principal Investigator — Mount Sinai Icahn School of Medicine
Locations (1):
- Light and Health Research Center, Menands, New York, United States

IPD SHARING:
Plan to Share IPD: No
Since this data collection occurs in a population with Alzheimer's disease, participants are generally not interested in individual results.